CLINICAL TRIAL: NCT06065475
Title: Ultrasound-guided Thyroid Cartilage Plane Block for Patients With Awake Tracheal Intubation: a Randomized Controlled Trial
Brief Title: Ultrasound-guided Thyroid Cartilage Plane Block for Awake Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tao Shan, Attending physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20230829-10
Record Dates: First submitted 2023-09-17; First posted 2023-10-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Superior Laryngeal Nerve Block
Keywords: Thyroid Cartilage; Superior Laryngeal Nerve; Difficult airway; ultrasound; Awake tracheal intubation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid Cartilage Plane Block Group (T Group) (Experimental): All patients received topical oral and pharyngeal anesthesia using 2.4% lidocaine spray. The pharyngeal surface was sprayed twice, with each spray lasting one second, and repeated after a 5-minute interval. Ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage plate as an anatomical landmark. 2.5ml of 2% lidocaine is injected on the surface of the thyroid cartilage each side. Subsequently, perform fiberoptic bronchoscope-guided subglottis and tracheal surface topical anesthesia using 5ml of 2% lidocaine. After completing surface anesthesia, perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.
  Interventions: Behavioral: Ultrasound-guided bilateral Thyroid Cartilage Plane Block
- the Control Group （C Group） (No Intervention): Patients in the C Group received topical oral and pharyngeal anesthesia using 2.4% lidocaine spray. The pharyngeal surface was sprayed twice, with each spray lasting one second, and repeated after a 5-minute interval. Patients in the C Group receive airway topical anesthesia using the fiberoptic bronchoscope-guided local anesthetic spray method throughout the vocal cord and tracheal with 5 ml 2% lidocaine respectively.

INTERVENTIONS:
Behavioral: Ultrasound-guided bilateral Thyroid Cartilage Plane Block — Use a SonoSite high-frequency linear array transducer (5-13 MHz, SonoSite, USA). Place the transducer parallel to the spine on one side of the neck, ensuring clear visualization of the thyroid cartilage plate under ultrasound. Employ ultrasound-guided out-of-plane techniques to display the needle insertion path and tip. Once the needle tip contacts the upper half of the thyroid cartilage plate, injecting 2.5ml of 2% lidocaine on the surface of the thyroid cartilage each side.
  Arms: Thyroid Cartilage Plane Block Group (T Group)

SUMMARY:
The goal of this clinical trial is to investigate the clinical effectiveness and safety of superior laryngeal nerve block through surface injection of local anesthetic solution on the thyroid cartilage in patients undergoing general anesthesia with endotracheal intubation. The main questions it aims to answer are the effectiveness of ultrasound-guided Thyroid Cartilage Plane Block for superior laryngeal nerve blockadethe and the safety and ease of performance.

All patients are divided into the Thyroid Cartilage Plane Block Group (T Group) and the Control Group (C Group). Patients in the C Group receive airway surface anesthesia using the fiberoptic bronchoscope-guided local anesthetic spray method throughout the procedure. In the experimental T Group, ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage as an anatomical landmark. Local anesthetic is injected on the surface of the thyroid cartilage.

Compare the following parameters between the two groups: duration of the blocking procedure, Ramsay Sedation Score, patient coughing upon contact of the fiberoptic bronchoscope with the vocal cords before intubation, comfort score immediately after intubation, and tracheal tube tolerance after successful intubation.

DETAILED DESCRIPTION:
Select 60 patients undergoing elective awake tracheal intubation surgery. Instruct patients to fast （no food or drink） for 8 hours before the procedure. Upon admission to the operating room, monitor patients' ECG （electrocardiogram）, BP （blood pressure）, and SpO2 （pulse oxygen saturation）. Establish intravenous access in the upper extremities and administer normal saline solution. Administer a loading dose of dexmedetomidine at 0.5 μg/kg over 5 minutes and remifentanil 0.5μg.kg-1, followed by an infusion at a rate of 0.3-0.6 μg/（kg·h） , 0.1μg.kg-1.min-1 by micropump infusion respectively. Perform radial artery puncture and catheter placement for invasive arterial pressure monitoring. Use a computer-generated random number table to allocate patients into two groups in a 1:1 ratio. To ensure objectivity, a nurse not involved in the study prepares sealed opaque envelopes containing the group assignments. All patients are divided into the Thyroid Cartilage Plane Block Group （T Group） and the Control Group （C Group）. All patients received topical oral and pharyngeal anesthesia using 2.4% lidocaine spray administered by an experienced anesthesiologist. The pharyngeal surface was sprayed twice, with each spray lasting one second, and repeated after a 5-minute interval. Each spray contained approximately 16 mg lidocaine. Patients in the C Group receive airway surface anesthesia using the fiberoptic bronchoscope-guided local anesthetic spray method throughout the vocal cord and tracheal with 5 ml 2% lidocaine respectively. In the experimental T Group, ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage plate as an anatomical landmark.2.5 ml 2% lidocaine local anesthetic is injected on the surface of the thyroid cartilage plate. The blocking procedure is as follows: Use a Sonosite high-frequency linear array transducer (5-13 MHz, Sonosite, USA). Place the transducer parallel to the spine on one side of the neck, ensuring clear visualization of the thyroid cartilage plate under ultrasound. Employ ultrasound-guided out-of-plane techniques to display the needle insertion path and tip. Once the needle tip contacts the upper half of the thyroid cartilage plate, inject 2.5ml of 2% lidocaine on the surface of the thyroid cartilage plate （the dosage is consistent with the commonly used local anesthetic volume for classic superior laryngeal nerve block methods in clinical practice）. Subsequently, perform fiberoptic bronchoscope-guided subglottic, and tracheal surface anesthesia. After completing surface anesthesia, select an appropriate-sized tracheal tube and perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for awake tracheal intubation surgery under general anesthesia.
2. Patients with difficult airways (e.g., limited cervical spine mobility, full stomach, partial airway obstruction, craniofacial deformities or trauma, micrognathia, mouth opening <3cm, Mallampati III or IV classification) posing challenges for mask ventilation or intubation.
3. Age between 18 and 65 years.
4. Gender is not restricted.
5. ASA classification of I or II.

Exclusion Criteria:

1. Cardiovascular dysfunction or arterial aneurysms.
2. Mental or neurological disorders or concomitant arterial aneurysms.
3. Infection at the puncture site.
4. Allergy to local anesthetics.
5. Continuous use of antiplatelet or anticoagulant medications preoperatively.
6. Hoarseness or coughing while drinking water.
7. Bronchial asthma.
8. Participation in other clinical trials within the previous 3 months before enrollment 9.r current participation in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
quality of airway anesthesia | Upon intubation
  TThe primary outcome in this trial was quality of airway anesthesia assessed on a 5-point scale,Quality of airway anesthesia was graded as: 0=no coughing or gagging in response to intubation, 1=mild coughing and/or gagging that did not hinder intubation, 2=moderate coughing and/or gagging that interfered minimally with intubation, 3=severe coughing and/or gagging that made intubation difficult and 4=very severe coughing and/or gagging that required additional local anesthetic and/or change in technique.The lower grade means a better quality of airway anesthesia.

SECONDARY OUTCOMES:
Mean Arterial Pressure （MAP） | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  Stable blood pressure indicates a good neural blockade effect.
Heart Rate （HR） | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  The smaller the heart rate fluctuations, the better the neural blockade effect.
Ramsay Sedation Score | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation
  The Ramsay Sedation Score is as follows: 6 points for unarousable, 5 points for slow response to stimulus, 4 points for asleep but easily aroused, 3 points for quiet and cooperative with orientation, 2 points for asleep, anxious, restless, and 1 point for asleep, agitated, and restless. Satisfactory sedation falls within 2-4 points, while oversedation is indicated by 5-6 points.
The number of patients with lowered pitch | Before intubation
  A lowered pitch indicates a good neural blockade effect.
The time of the block procedure | From ultrasound probe positioning the target to completion of drug administration
  The neural blockade procedure time reflects the ease of the operation, with a shorter time indicating a simpler neural blockade procedure.
Record coughing in patients when the fiberoptic bronchoscope touches the glottis | Before intubation
  The patient's coughing upon contact of the fiberoptic bronchoscope with the vocal cords before intubation reflects the effectiveness of neural blockade. A lower degree of coughing indicates a better neural blockade effect. 1 point for no response, 2 points for mild cough, 3 points for severe cough.
The tolerance of the tube | After successful intubation
  The tolerance of the tube reflects the patient's tolerance to awake tracheal intubation. A higher level of tolerance indicates a better neural blockade effect. 3 points for severe resistance requiring immediate general anesthesia, 2 points for restlessness and mild resistance, 1 point for cooperation.
Adverse reactions such as coughing and nausea/ vomiting.. | During intubation
  The lower the incidence of coughing, nausea, and vomiting, the better the neural blockade effect.
Occurrences of sore throat and lowered pitch | Post-extubation,24 hours after surgery
  Pharyngeal pain and decreased vocal tone are used to assess postoperative complications of neural blockade.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shan, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiles JR, Kelly J, Mostafa SM. Hypotension and bradycardia following superior laryngeal nerve block. Br J Anaesth. 1989 Jul;63(1):125-7. doi: 10.1093/bja/63.1.125. PMID 2765339
- [Background] Canty DJ, Poon L. Superior laryngeal nerve block: an anatomical study comparing two techniques. J Clin Anesth. 2014 Nov;26(7):517-22. doi: 10.1016/j.jclinane.2014.03.005. Epub 2014 Oct 16. PMID 25439414
- [Background] Fowler JG, VanEenenaam DP Jr, Johnson KN, Courtemanche CD, Strathman AJ, Reynolds JE. Single midline injection for bilateral superior laryngeal nerve block. J Clin Anesth. 2020 Nov;66:109922. doi: 10.1016/j.jclinane.2020.109922. Epub 2020 Jun 6. No abstract available. PMID 32516680

DOCUMENTS (1):
  • Study Protocol (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT06065475/Prot_000.pdf